CLINICAL TRIAL: NCT05014425
Title: Risk Factors Predicting Development of Pancreatic Fistula Following Pancreaticoduodenectomy
Brief Title: Risk Factors for Post Whipple Pancreatic Fistula
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy A. Hassan, Dr., Assiut University
Other Study IDs: Pancreatic fistula
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreaticoduodenectomy

SUMMARY:
Postoperative pancreatic fistula (POPF) following pancreaticoduodenectomy is considered a life-threatening complication. This study was designed to analyze the risk factors for development of such fistula in a tertiary care center (Al-Rajhi Liver Hospital/ Assiut University).

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent pancreaticoduodenectomy for pancreatic cancer

Exclusion Criteria:

* All types of pancreatic resection other than pancreaticoduodenectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients underwent pancreaticoduodenectomy at Al-Rajhi liver Hospital, Assiut university from January 2017 to December 2020
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Development of pancreatic fistula following pancreaticoduodenectomy | Baseline
  Analysis of risk factors for development of pancreatic fistula following pancreaticoduodenectomy